CLINICAL TRIAL: NCT06003387
Title: Phase 3b, Open-label, Multicenter, Single-dose Study Investigating Efficacy and Safety of CSL222 (Etranacogene Dezaparvovec) Gene Therapy Administered to Adult Subjects With Severe or Moderately Severe Hemophilia B With Detectable Pretreatment AAV5 Neutralizing Antibodies
Brief Title: Efficacy and Safety of CSL222 (Etranacogene Dezaparvovec) Gene Therapy in Adults With Hemophilia B With Pretreatment Adeno-associated Virus Serotype 5 (AAV5) Neutralizing Antibodies (Nabs)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSL222_3005; 2023-509590-23-00 (EU CTIS Number)
Record Dates: First submitted 2023-08-01; First posted 2023-08-22 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-08

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CSL222 (Experimental): Participants will receive CSL222 as a single intravenous (IV) infusion of 2 × 10^13 genome copies per kilogram (gc/kg) on Day 1.
  Interventions: Genetic: CSL222 (AAV5-hFIXco-Padua)

INTERVENTIONS:
Genetic: CSL222 (AAV5-hFIXco-Padua) — Administered as a single IV infusion.
  Other Names: Etranacogene dezaparvovec

SUMMARY:
The purpose of this study is to assess the risk of bleeding due to failure of expected pharmacological action of CSL222 in adults with severe or moderately severe hemophilia B with detectable pretreatment AAV5 Nabs.

ELIGIBILITY:
Inclusion Criteria:

* nd considered legally an adult, as defined by country regulations.
* •Has congenital hemophilia B with known severe or moderately severe FIX deficiency (less than or equal to [<=] 2% of normal circulating FIX) for which the participant is on continuous routine FIX prophylaxis.
* • Has 2 consecutive detectable AAV5 NAb titer results between Screening and Visit L-Final using a validated AAV5 NAb assay (based on central laboratory results).
* • Has greater than (>) 150 previous exposure days to FIX replacement therapy.
* • Has been on stable FIX prophylaxis for at least 2 months before Screening.
* • Has demonstrated capability to independently, accurately, and in a timely manner complete the eDiary during the Lead-in Period, as judged by the investigator.
* • Acceptance to adhere to contraception guidelines.
* • Able to provide informed consent after receipt of verbal and written information about the study.
* • Investigator believes that the participant (or the participant's legally acceptable representative[s]) understands the nature, scope, and possible consequences of the study and is able to adhere to the study procedures.

Exclusion Criteria:

* • History of FIX inhibitors or positive FIX inhibitor test at Prescreening, Screening or Visit L-Final (based on central laboratory results).
* • Screening or Visit L-Final laboratory values (based on central laboratory results) of total bilirubin > 2 × the upper limit of normal (ULN) (except if caused by Gilbert's syndrome).
* • Screening or Visit L-Final laboratory values (based on central laboratory results) of any of the following laboratory abnormalities:
* a) ALT > 2 × the ULN
* b) AST > 2 × the ULN
* c) Alkaline phosphatase > 2 × the ULN
* d) Serum creatinine > 2 × the ULN
* e) Hemoglobin less than (<) 8 g/dL
* • Any condition other than hemophilia B resulting in an increased bleeding tendency.
* • Thrombocytopenia, defined as a platelet count <50 × 10^9/L, at Screening or Visit L Final (based on central laboratory results).
* • Any uncontrolled or untreated infection (human immunodeficiency virus [HIV], hepatitis B virus [HBV] and hepatitis C virus [HCV], or any other significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, cardiovascular, hematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease, alcoholism, drug dependency, or any other psychological disorder evaluated by the investigator to interfere with adherence to the clinical study protocol procedures or with the degree of tolerance to CSL222.
* • Known history of allergy to corticosteroids or known medical condition that would require chronic administration of oral corticosteroids.
* • Known uncontrolled allergic conditions or allergy / hypersensitivity to any component of the CSL222 excipients (ie, sucrose, potassium chloride, potassium dihydrogen phosphate, sodium chloride, and disodium hydrogen phosphate).
* • Previous AAV5 gene therapy treatment.
* • Receipt of an experimental agent or device within 60 days before Screening until the end of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2028-10-04 (Estimated); Study Completion 2032-04-02 (Estimated)

PRIMARY OUTCOMES:
Annualized Bleeding Rate (ABR) | Months 7 to 18 after CSL222 treatment
  The total bleeding episodes will be analyzed. ABR is calculated as the total bleeding episodes divided by the total time at risk.

SECONDARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events (TEAEs) | Up to 60 months after CSL222 treatment
Percentage of participants with TEAEs | Up to 60 months after CSL222 treatment
Number of TEAEs | Up to 60 months after CSL222 treatment
Change in Liver ultrasound | Up to 60 months after CSL222 treatment
Number of participants who develop Factor IX (FIX) Inhibitors | Up to 60 months after CSL222 treatment
Percentage of participants who develop FIX Inhibitors | Up to 60 months after CSL222 treatment
Change in hematology and biochemistry parameters | Up to 60 months after CSL222 treatment
Number of participants with clinically significant increase in Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) | Up to 60 months after CSL222 treatment
Percentage of participants with clinically significant increase in ALT or AST | Up to 60 months after CSL222 treatment
Corticosteroid use for ALT or AST increases after CSL222 treatment | Up to 60 months after CSL222 treatment
Number of participants with clinically significant Alpha-fetoprotein (AFP) | Baseline and up to 60 months after CSL222 treatment
Percentage of participants with clinically significant AFP | Baseline and up to 60 months after CSL222 treatment
Number of participants with infusion related reactions or hypersensitivity reactions | Throughout CSL222 infusion period and up to 60 months after CSL222 treatment
Percentage of participants with infusion related reactions or hypersensitivity reactions | Throughout CSL222 infusion period and up to 60 months after CSL222 treatment
Change in the Uncontaminated Endogenous FIX activity | Baseline and up to Months 6, 12, and 18 after CSL222 treatment
Annualized consumption of FIX replacement therapy | Months 7 to 18 after CSL222 treatment
Annualized infusion rate of FIX replacement therapy | Months 7 to 18 after CSL222 treatment
Number of participants remaining free of continuous FIX prophylaxis | Months 7 to 18 after CSL222 treatment
Percentage of participants remaining free of continuous FIX prophylaxis | Months 7 to 18 after CSL222 treatment
ABR for spontaneous bleeding episodes | Months 7 to 18 after CSL222 treatment
ABR for joint bleeding episodes | Months 7 to 18 after CSL222 treatment
ABR for FIX-treated bleeding episodes | Months 7 to 18 after CSL222 treatment
Correlation analysis of FIX activity levels with baseline AAV5 NAb titers | Months 7 to 18 after CSL222 treatment
Number of participants with new target joints and resolved pre-existing target joints | Months 7 to 18 after CSL222 treatment
  Target joint is defined as 3 or more spontaneous bleeding episodes into a single joint.
Number of participants with zero bleeding episodes and zero FIX-treated bleeding episodes | Months 7 to 18 after CSL222 treatment
Percentage of participants with zero bleeding episodes and zero FIX-treated bleeding episodes | Months 7 to 18 after CSL222 treatment
Change in the EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) Visual Analogue Scale (VAS) Overall Score | Baseline and up to 18 months after CSL222 treatment
  The EQ-5D-5L questionnaire visual analogue scale (VAS) measures overall health status on a vertical VAS ranging from 0 to 100. A higher score indicates better quality of life. The change from baseline in the EQ-5D-5L VAS score will be determined.
Change in the EQ-5D-5L Index Scores | Baseline and up to 18 months after CSL222 treatment
  The EQ-5D-5L questionnaire descriptive system of health-related quality of life consists of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) for which responses will be recorded on 5 levels of severity (no problems, slight problems, moderate problems, severe problems, and extreme problems). The responses will be converted into a single index utility score (typically between -0.6 and 1). A higher score indicates better quality of life. The change from baseline in the EQ-5D-5L index score will be determined.
Number of Participants with Uncontaminated Endogenous FIX Activity of Greater than or Equal to (>=) 5% | Months 7 to 18 after CSL222 treatment
Percentage of Participants with Uncontaminated Endogenous FIX Activity of >= 5% | Months 7 to 18 after CSL222 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (25):
- United States (2):
  - University of California, San Diego (UCSD) - 84000460, San Diego, California
  - University of Michigan - 84000285, Ann Arbor, Michigan
- Australia (4):
  - Royal Prince Alfred Hospital - 03600044, Camperdown, New South Wales
  - Royal Brisbane Hospital - 03600045, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital - 03600043, Melbourne, Victoria
- McMaster University - Hamilton - 12400017, Hamilton, Ontario, Canada
- Hong Kong (2):
  - Queen Mary Hospital - 34400001, Hong Kong
  - Prince of Wales Hospital Chinese University of Hong Kong - 34400002, Shatin
- Sheba Medical Center - 37600004, Tel Litwinsky, Israel
- Centro de Investigacion Clinica GRAMEL S.C. - 48400003, Mexico City, Mexico City, Mexico
- King Faisal Specialist Hospital and Research Center - 68200001, Riyadh, Saudi Arabia
- National University Hospital - 70200002, Singapore, Singapore
- Haemophilia Comprehensive Care Centre - 71000001, Johannesburg, South Africa
- South Korea (3):
  - Kyungpook National University Hospital - 41000014, Daegu
  - Kyung Hee University Hospital at Gangdong - 41000015, Seoul
  - Severance Hospital, Yonsei University Health System - 41000013, Seoul
- Taiwan (5):
  - Tri-Service General Hospital - 15800012, Taipei, Neihu District
  - Kaohsiung Medical University Chung-Ho Memorial Hospital (KMUH) - 15800011, Kaohsiung City, Sanmin District
  - Changhua Christian Hospital (CCH) - 15800009, Chang-hua
  - Taichung Veterans General Hospital - 15800007, Taichung
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (3):
  - Ege University Medical Faculty - 79200002, Bornova
  - Gaziantep University Sahinbey Research and Practice Hospital - 79200004, Gaziantep
  - Özel Acibadem Adana Hastanesi - 79200003, Seyhan

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (ie FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.